CLINICAL TRIAL: NCT00215748
Title: Feasibility of A Reduced Dexamethasone Pre-Medication Dose in Elderly Patients Treated With Weekly Docetaxel
Brief Title: Reduced Dexamethasone Pre-Medication Dose in Elderly Patients Receiving Weekly Docetaxel
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Geriatric Oncology Consortium (Other)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOC S-010
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Breast Cancer; Lung Cancer
Keywords: Elderly; Weekly
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms | interventions — Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone

SUMMARY:
This study is to explore the feasibility of an alternative dose of dexamethasone pre-medication in older breast and lung cancer patients who are receiving weekly docetaxel chemotherapy.

DETAILED DESCRIPTION:
Dose-limiting edema and effusions associated with cumulative docetaxel administraton have necessitated the recommendation that all patients should be premedicated with oral corticosteroids such as dexamethasone prior to docetaxel administration. Dexamethasone pre-medication may also decrease the incidence and severity of acute hypersensitivity reactions associated with docetaxel administration. However, administration of weekly dexamethasone can cause additional untoward side effects, especially in the older population. If the data from this phase II study is encouraging, a study to evaluate an even lower dose of dexamethasone can be conducted.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65 years;
* breast or lung cancer patients to receive docetaxel therapy as per protocol;
* corticosteroid administration, other than what is prescribed in this protocol, is not permitted during study participation, except topical administration and for adverse events;
* performance status ECOG 0-2;
* peripheral neuropathy ≤ 1;
* adequate kidney and liver functions
* signed study-specific informed consent

Exclusion Criteria:

* Patients who have received an investigational drug within 4 weeks of registration;
* Prior or concurrent malignancies (other than surgically treated carcinoma in situ;
* Serious medical or psychiatric illness which would prevent informed consent;
* Life expectancy < 3 months;
* Active uncontrolled bacterial, viral, or fungal infection until these conditions are corrected or controlled.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-08; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of a reduced dexamethasone pre-medication dose in elderly lung and breast cancer patients receiving weekly docetaxel therapy with respect to incidence of: Grade 3/4 fluid retention
Grade 3/4 hypersensitivity

SECONDARY OUTCOMES:
To evaluate the incidence of toxicity of a reduced dexamethasone pre-medication dose in elderly lung and breast cancer patients receiving weekly docetaxel with respect to: fluid retention (all grades)
hypersensitivity (all grades)

CONTACTS AND LOCATIONS:
Overall Officials: William Ershler, MD, Principal Investigator — Geriatric Oncology Consortium
Locations (1):
- Baltimore, Maryland, United States

REFERENCES:
- See also: Geriatric Oncology Consortium website — http://www.thegoc.org